CLINICAL TRIAL: NCT04899219
Title: An Open-label, Single-dose Study to Investigate the Pharmacokinetics of ACT-1014-6470 in Subjects With Severe Renal Impairment Compared to Control Subjects
Brief Title: A Study to Investigate the Pharmacokinetics of ACT-1014-6470 in Subjects With Severe Renal Impairment Compared to Control Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ID-087-104
Record Dates: First submitted 2021-05-19; First posted 2021-05-24 (Actual); Last update posted 2021-11-29 (Actual); Status verified 2021-11

CONDITIONS: Healthy
MeSH Terms: interventions — ACT-1014-6470

STUDY DESIGN:
Intervention Model Description: This is a prospective, open-label, single-dose, parallel-group, Phase 1 study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (subjects with severe renal impairment) (Experimental)
  Interventions: Drug: ACT-1014-6470 40 mg
- Group B (control subjects) (Experimental)
  Interventions: Drug: ACT-1014-6470 40 mg

INTERVENTIONS:
Drug: ACT-1014-6470 40 mg — ACT-1014-6470 will be available as soft gelatin capsules for oral administration formulated at a dose strength of 20 mg.

SUMMARY:
An open-label, single-dose study to investigate the pharmacokinetics of ACT-1014-6470 in subjects with severe renal impairment compared to control subjects

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent in a language understandable to the subject prior to any study-mandated procedure.
* Male or female subject aged at least 18 years at Screening.
* Women of non-childbearing potential (e.g. post-menopausal)

Additional inclusion criteria for subjects with severe renal impairment (Group A).

- Severe renal function impairment as confirmed at Screening based on an estimated glomerular filtration rate (eGFR) using the Modification of Diet in Renal Disease (MDRD) formula of < 30 mL/min (not on dialysis).

Additional inclusion criteria for control subjects (Group B):

* Normal renal function as confirmed at Screening based on eGFR.
* Each control subject must be matched to the values of one subject with severe renal impairment based on age (±10 years difference allowed), BMI (±15% difference allowed), and sex, determined by results at Screening.

Exclusion Criteria:

- Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-06-16 (Actual); Primary Completion 2021-11-12 (Actual); Study Completion 2021-11-12 (Actual)

PRIMARY OUTCOMES:
PK of ACT-1014-6470 - Cmax | Blood samples for PK analysis will be drawn at various time points (total duration: up to 6 days in Group A, up to 4 days in Group B).
  For both Group A (subjects with severe renal impairment) and Group B (control subjects)

OTHER OUTCOMES:
PK of ACT-1014-6470 - Tmax | Blood samples for PK analysis will be drawn at various time points (total duration: up to 6 days in Group A, up to 4 days in Group B).
  For both Group A (subjects with severe renal impairment) and Group B (control subjects)
Group B (control subjects): PK of ACT-1014-6470 - AUC0-inf | Blood samples for PK analysis will be drawn at various time points (total duration: up to 6 days in Group A, up to 4 days in Group B).
  For both Group A (subjects with severe renal impairment) and Group B (control subjects)
Group B (control subjects): PK of ACT-1014-6470 - T1/2 | Blood samples for PK analysis will be drawn at various time points (total duration: up to 6 days in Group A, up to 4 days in Group B).
  For both Group A (subjects with severe renal impairment) and Group B (control subjects)

CONTACTS AND LOCATIONS:
Locations (1):
- APEX GmbH, Munich, Germany

IPD SHARING:
Plan to Share IPD: No